CLINICAL TRIAL: NCT05999682
Title: Improvement of Organ Function by Apigenin in Elderly Patients With Sepsis: A Single-center, Single-blind, Randomized, Placebo-controlled, Pilot Clinical Trial
Brief Title: Improvement of Organ Function by Apigenin in Elderly Patients With Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Director of the department of critical care medicine, Principal Investigator, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-KY-085-03
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; apigenin; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Apigenin

STUDY DESIGN:
Intervention Model Description: Treatment group: Intragastric tube injection of ground apigenin tablet 50 mg with 5 ml of sterilized water + conventional standardized treatment, for 4 days or ICU discharge.
  Control group: Intragastric tube injection of 5 ml of sterilized water + conventional standardized treatment, for 4 days or ICU discharge.
Who Masked: Participant
Masking Description: Single(Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apigenin (Experimental): Intragastric tube injection of ground apigenin tablet 50 mg with 5 ml of sterilized water + conventional standardized treatment, for 4 consecutive days.
  Interventions: Other: apigenin
- sterilized water (Placebo Comparator): Gastric tube injection of 5 ml of sterilized water for injection + conventional standardized treatment, for 4 consecutive days.
  Interventions: Other: sterilized water

INTERVENTIONS:
Other: apigenin — Intragastric tube injection of ground apigenin tablet 50 mg with 5 ml of sterilized water + conventional standardized treatment, for 4 consecutive days.
  Arms: apigenin
Other: sterilized water — Intragastric tube injection of 5 ml of sterilized water + conventional standardized treatment, for 4 consecutive days.
  Arms: sterilized water

SUMMARY:
In this single-center, randomized, single-blind, placebo-controlled pilot clinical trial. The effect of apigenin on the improvement of organ function will be investigated in elderly patients with sepsis. Researchers will screen patients admitted to the Department of Critical Care Medicine at Zhujiang Hospital to identify patients with sepsis based on including and excluding criteria and obtain informed consent and randomize them into groups. The treatment group will be given apigenin tablets 50mg ground with 5ml of sterilized water for intra-gastric tube injection; the control group will be given an equal volume of sterilized water for intra-gastric tube injection. The changes in SOFA score and other clinically meaningful outcomes in 4 days will be collected.

DETAILED DESCRIPTION:
Investigational drug: Apigenin Study title: Improvement of Organ function by Apigenin in Elderly Patients With Sepsis: A Single-center, Single-blind, Randomized, Placebo-controlled, pilot Clinical Trial Principal Investigator: Zhanguo Liu, professor, Department of Critical Care Medicine, Zhujiang Hospital, Southern Medical University Study subjects: Elderly septic/septic shock patients who meet the diagnostic criteria of the 2016 International Sepsis Guidelines.

Study objectives: The objective of the study is to determine whether apigenin, compared to placebo, improves organ dysfunction scores (SOFA scores) in elderly septic patients.

Study design: A single-center, single-blind, randomized, placebo-controlled pilot Clinical Trial.

Method: Apigenin group: Intragastric tube injection of ground apigenin tablet 50 mg with 5 ml of sterilized water + conventional standardized treatment, for 4 days or until ICU discharge. Placebo control group: Gastric tube injection of 5 ml of sterilized water for injection + conventional standardized treatment, for 4 days or ICU discharge.

Course: 4 days Sample size: 20 The number of study center: 1

Study center:

1. Department of Critical Care Medicine of Zhujiang Hospital, Guangzhou, Guangdong, China Primary endpoint: 96-hour Sequential Organ Failure Assessment (SOFA) score

   Secondary endpoints:
2. The state of inflammatory response: the serum level of interleukin-6(IL-6) and C-reactive protein (CRP) at 96 h after randomization.
3. The state of liver function: the serum level of transaminase (AST#ALT) #total bilirubin at 96 h after randomization.
4. The state of lung function: oxygenation index (PaO2/FiO2) at 96h after Randomization.
5. The state of kidney function: the serum level of Creatinine (Cr)#blood urea nitrogen (BUN)# at 96 h after randomization.
6. The state of infection: the serum level of procalcitonin (PCT) at 96 h after randomization.
7. The state of circulation system: the serum level of lactate at 96 h after Randomization.
8. The duration of successful cessation of supportive therapies for organ dysfunction including vasoactive agents, mechanical ventilation.
9. The daily urine output#duration of continuous renal replacement therapy (CRRT) #fluid balance.
10. The length of stay in ICU.

Safety endpoints:

1. adverse events
2. Serious adverse events

ELIGIBILITY:
Inclusion Criteria:

1. age ≥65 years;
2. meeting the diagnostic criteria of the 2016 International Sepsis Guidelines;
3. subjects who voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

1. patients who are allergic to the study products;
2. patients who are unable to feed via gastrointestinal nutrition tube.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
96-hour Sequential Organ Failure Assessment (SOFA) score | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  The SOFA score is the Sequential Organ Failure Score, which is used to assess a patient's prognosis by determining the degree of impairment of major organ function. The score is divided into 6 sections: respiratory, coagulation, hepatic, cardiovascular, central nervous system, and renal, and ranges from 0 to 4, with higher SOFA scores associated with a higher incidence of poor prognosis.

SECONDARY OUTCOMES:
inflammatory response(1) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of C-reactive protein(CRP)
inflammatory response(2) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of interleukin-6(IL-6)
Duration of use of vasoactive drugs | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  The duration from the vasoactive drugs administration to the successful cessation in hours( The successful cessation is defined as the attainment of a clinician-prescribed mean arterial pressure target for more than 24-hours without the use of vasoactive drugs.This outcome measure is intended only for patients receiving vasoactive drugs)
liver function(1) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of Alanine transaminase(ALT)
liver function(2) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of Aspartate transaminase (AST)
liver function(3) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of total bilirubin(TBil)
lung function | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  oxygenation index(PaO2/FiO2),the patients treated with extracorporeal membrane oxygenation will not collect this indicator
kidney function(1) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  serum level of Creatinine (Cr)
kidney function(2) | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  serum level of blood urea nitrogen(BUN)
Indicators of infection | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of procalcitonin(PCT)
The level of lactate | The outcome will be assessed at the 0,1,2,3,4 day after enrollment
  the serum level of lactic acid
The Duration of use of mechanical ventilation (MV) | The outcome will be assessed at the 28 day after enrollment
  The duration from the MV administration to the successful cessation in hours( The successful cessation is defined as the termination of MV for more than 48-hours. This outcome measure is intended only for patients receiving MV)
The duration of CRRT | The outcome will be assessed at the 28 day after enrollment
  The duration of CRRT therapy in hours
Daily urine output | The outcome will be assessed at the 1,2,3,4 day after enrollment
  Daily urine output in milliliters from 0:00 - 24:00
fluid balance | The outcome will be assessed at the 1,2,3,4 day after enrollment
  Net fluid intake and output in 24 hours
The length of ICU stay | The outcome will be assessed at the 28 day after enrollment
  ICU length of ICU stay

OTHER OUTCOMES:
Incidence of adverse events | The outcome will be assessed at the 28 day after enrollment
  A adverse event refers to any adverse medical event that occur after the intervention of trial. The adverse events are not necessarily causally related to the trial treatment.
Incidence of serious adverse events | The outcome will be assessed at the 28 day after enrollment
  Any adverse medical event occurs at any dose that meets one or more of the following criteria: 1. causes death 2.life-threatening 3. requires hospitalization or hospitalization for an extended period of time 4. causes permanent or significant disability and functional defects 5. causes deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Liu, M.D.PhD, Principal Investigator — Department of Critical Care Medicine of Zhujiang Hospital
Locations (1):
- Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and analyzed during the study are available from the corresponding author on reasonable request.